CLINICAL TRIAL: NCT00892944
Title: An Open Label Positron Emission Tomography (PET) Study With [11C]AZ12713580 to Determine Central mGluR5 Receptor Occupancy of AZD2516 After Oral Administration to Healthy Subjects
Brief Title: An Open Label Positron Emission Tomography (PET) Study to Determine Central mGluR5 Receptor Occupancy of AZD2516
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D2080C00009
Record Dates: First submitted 2009-04-28; First posted 2009-05-05 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: Positron Emission Tomography; Phase 1; Healthy volunteers; AZD2516

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD2516
  Interventions: Drug: AZD2516

INTERVENTIONS:
Drug: AZD2516 — Fractionated single oral dose

SUMMARY:
The purpose of this study is to determine if AZD2516 binds to mGluR5 receptors in the brain. This will then help to make accurate predictions of efficacy and dosing in the future development programme.

ELIGIBILITY:
Inclusion Criteria:

* Normal MRI scan
* Healthy male or non-fertile females
* Body Mass Index (BMI) of ≥19 to ≤28 kg/m2 and weight of ≥50 to ≤100 kg

Exclusion Criteria:

* History of disease or condition that may interfere with the objectives of the study
* History of previous or ongoing psychiatric disease/condition
* Concomitant medication

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2009-04; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography to determine if AZD2516 can displace the radioligand [11C]AZ12713580 and describe relationship between AZD2516 exposure and mGluR5 receptor occupancy | 1 Month: Baseline and 3 PET examinations

SECONDARY OUTCOMES:
Safety and tolerability of AZD2516 by adverse events, vitals signs, ECG, body temperature and laboratory variables | Assessed at each visit from baseline to follow-up visit
To investigate the Pharmacokinetics of AZD2516 | 1 Month: 3 doses AZD2516 and 16 planned PK samples after each dose

CONTACTS AND LOCATIONS:
Overall Officials: Ingemar Bylesjo, MD, PhD, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Stockholm, Sweden; Michael O'Malley, Study Director — AstraZeneca R&D, Södertälje, Sweden
Locations (1):
- Research Site, Stockholm, Sweden